CLINICAL TRIAL: NCT03975504
Title: Community-based Lung Cancer Screening With Low-dose CT in China (CLUS Study) Version 2.0
Brief Title: China Lung Cancer Screening (CLUS) Study Version 2.0
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Baohui Han, Director, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CHEST1809
Record Dates: First submitted 2019-06-04; First posted 2019-06-05 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms | interventions — Tomography, X-Ray Computed; Optical Imaging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LDCT Screening (Other): LDCT was performed at baseline + 2 biennial repeated LDCT rounds
  Interventions: Device: Low Dose Computed Tomography; Device: artificial intelligence (AI); Diagnostic Test: autofluorescence imaging (AFI)

INTERVENTIONS:
Device: Low Dose Computed Tomography — LDCT were performed in screening arm. The abnormal nodules were defined as noncalcified nodules (NCN) larger than 5 mm
Device: artificial intelligence (AI) — AI was performed in high-risk individuals recruitment and lung nodules management
Diagnostic Test: autofluorescence imaging (AFI) — AFI applied in screening of centrally located SCC.

SUMMARY:
Our previous study, china lung cancer screening study version 1.0, had proven that LDCT led to a 74.1% increase in detecting early-stage lung cancer compare to usual care (NCT02898441). The present one arm study is performed to evaluate the efficacy of new techniques in improving the implementation of lung cancer screening and validate our previous findings. 6000 high-risk subjects (age 45-75) were recruited to take LDCT screening. (Baseline + 2 biennial repeated LDCT screening). Follow-up for lung cancer incidence, lung cancer mortality and overall mortality was performed. Blood samples were stored in a Biobank. Management of positive screening test was carried out by a pre-specified protocol.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants were those aged 45-75 years, and with either of the following risk factors:

  1. history of cigarette smoking ≥ 20 pack-years, and, if former smokers, had quit within the previous 15 years;
  2. malignant tumors history in immediate family members;
  3. personal cancer history;
  4. professional exposure to carcinogens;
  5. long term exposure to second-hand smoke;
  6. long term exposure to cooking oil fumes.

Exclusion Criteria:

1. Had a CT scan of chest within last 12 months
2. History of any cancer within 5 years

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
The mortality rate of lung cancer | 5 years
  Assess lung cancer mortality within next 5 years after first round of screening
The attendance rate of high-risk individuals | 5 year
  Evaluate the ability of AI in enhancing the attendance rate of high-risk individuals
Diagnostic accuracy rate of lung cancer | 5 year
  Evaluate the ability of AI, AFI and molecular biomarkers in enhancing the diagnostic accuracy rate of lung cancer

SECONDARY OUTCOMES:
The mortality of all-cause | 5 years
  Assess all-cause mortality within next 5 years after first round of screening
The detection rate of lung nodules | 5 year
  Assess lung nodules detection rate, and the types and sizes of nodules detected in LDCT screening
The incidence rate lung cancer | 5 years
  Assess the number of lung cancer incidences after each round of screening

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang Y, Liu W, Zhang H, Sun B, Chen T, Hu M, Zhou H, Cao Y, Han B, Wu L. Extracellular vesicle long RNA markers of early-stage lung adenocarcinoma. Int J Cancer. 2023 Apr 1;152(7):1490-1500. doi: 10.1002/ijc.34386. Epub 2022 Dec 15. PMID 36451312